CLINICAL TRIAL: NCT05286086
Title: Randomized Controlled Trial Comparing the Effect of a Multimodal Prehabilitation Program During Neoadjuvant Treatment Versus a Multimodal Prehabilitation After Neoadjuvant Treatment for Patients Undergoing Resection of Rectal Cancer.
Brief Title: Prehabilitation in Rectal Cancer: During Neoadjuvant Therapy vs Preoperative
Acronym: PREHAREC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Laura Mora-Lopez, PhD, MD, Colorrectal Surgeon, Associate Professor, Corporacion Parc Tauli
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PREHAREC
Record Dates: First submitted 2022-02-09; First posted 2022-03-18 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Rectal Cancer, Adenocarcinoma; Chemoradiotherapy
Keywords: RECTAL CANCER; PREAHBILITATION; NEOADJUVANCY; COMPREHENSION COMPLICATION INDEX
MeSH Terms: conditions — Rectal Neoplasms | interventions — Preoperative Exercise

STUDY DESIGN:
Intervention Model Description: Prospective , unicentric, randomized
Masking Description: due to the characteristics of the study, it is not possible to perform masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PREHAB-PREOP (Sham Comparator): PREHABILITATION BEFORE SURGERY
  Interventions: Behavioral: prehabilitation
- PREHAB-NEOADJ (Experimental): PREHABILITATION DURING NEOADJUVANCY AND BEFORE SURGERY
  Interventions: Behavioral: prehabilitation

INTERVENTIONS:
Behavioral: prehabilitation — Control of the physical, nutritional and psychological preparation of the patient who will undergo rectal cancer surgery

SUMMARY:
Control of the effect of prehabilitation on postoperative morbidity, assessed by the Comprehensive Complication Index (CCI), in patients diagnosed with rectal cancer that will receive neoadjuvant Quimiorradiotherapy (NCRT) and subsequent surgery, performed at the beginning of NCRT or before surgery.

DETAILED DESCRIPTION:
According to the annual report of the Spanish Medical Oncology Association (SEOM), in Spain and without differentiating by sex, colorectal cancer will be the cancer with the highest incidence by 2021; with 43.581 new cases estimated for such year, 14.209 of these will be of rectal cancer. In rectal cancer, surgery remains the cornerstone; however, it is already known that local recurrences are frequent. That is why one of the main milestones rectal cancer treatment, is the multimodal therapy approach. It consists of implementing a neoadjuvant chemoradiotherapy treatment (NCRT) prior to surgical intervention. With this, local control of the disease is achieved, metastases are reduced have resulted in a five-year survival. Subsequently, depending on the definitive pathological results, patients should also complete treatment with postoperative chemotherapy. It is known that patients undergoing neoadjuvant treatment experience a wide variety of side effects, which can cause loss of muscle and cardiovascular function, loss of their functional capacity and increased fatigue. This worsens the quality of life of the patient and can sometimes cause the interruption of neoadjuvant treatment and have repercussions on the prognosis. Not only do these side effects affect the course of neoadjuvant treatment, but also declines the physiological reserve, making the patient arrive in sub-optimal conditions for surgery. This has an impact on postoperative morbidity and mortality, and secondarily, in the increase of hospital stay.

The concept of functional capacity appears ¨as the nutritional, physical and emotional state that a person has to face a stressful situation, such as surgical treatment. It is believed that if functional capacity is enhanced, postoperative morbidity can be reduced and the patient's recovery can also be improved. That is why trimodal programs are created, specifically selected for their potential cumulative or synergistic effects on health outcomes to prepare patients to face surgery at all three levels. These programs are known as prehabilitation.

Currently there are studies that show that prehabilitation improves the results of patients who must undergo different major surgical procedures, among them in colorectal surgery. Our group has recently presented a study that shows that trimodal prehabilitation contributes to reducing postoperative morbidity and overall hospital stay in patients operated on for colorectal neoplasia. There are also systematic reviews that conclude that prehabilitated patients who must undergo major surgery (speaking of 435 patients and 9 studies) present a decrease in the incidence of major postoperative complications. On the other hand, there are studies that show that prehabilitation in patients who must receive neoadjuvant therapy reduces the decrease of functional capacity that treatment produces on patients. As also shown by the Rex Trial, a randomized study on 48 patients. In an attempt to unite the two lines start the study, it will be a novel one , with only two previously published studies in this area. The intention is demonstrate that when prehabilitation is started before commencing neoadjuvant therapy in patients who are diagnosed with rectal cancer and who are subject to neoadjuvant therapy, will reduce the effect on functional capacity, and that patients will present less postoperative morbidity and better postoperative recovery.

ELIGIBILITY:
Inclusion Criteria:

* Patient with rectal tumour and selected to initiate NRCT
* Patient must know the study and sign informed consent.
* Patient must accept the conditions necessaries to carry out the prehabilitation.

Exclusion Criteria:

* Refusal of the patient to sign the informed consent.
* Baseline pathology that makes it impossible to carry out prehabilitation.
* Progression of the disease during the study period.
* Emergency surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Comprehension Complication Index (CCI) | through study completion, an average of 1 yea
  Morbidity after surgery of rectal cancer: CCI - value 0-100

SECONDARY OUTCOMES:
6 minutes walking test (6MWT) | through study completion, an average of 1 yea
  Walking test that helps calculation of the number of daily steps to be carried out (5.000 to 10.000) daily steps
Hospital Anxiety and Depression Scale (HADS) test : anxious and depresion scale | through study completion, an average of 1 yea
  Calculation of level of anxiety or depression in mild, moderate or severe. Allows referral of the patient to the psychology service

CONTACTS AND LOCATIONS:
Overall Officials: Laura Mora, Dr, Principal Investigator — Parc Tauli University Hospital
Locations (1):
- Laura Mora López, Sabadell, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Berho M, Narang R, Van Koughnett JA, Wexner SD. Modern multidisciplinary perioperative management of rectal cancer. JAMA Surg. 2015 Mar 1;150(3):260-6. doi: 10.1001/jamasurg.2014.2887. PMID 25629513
- [Result] Herman JM, Narang AK, Griffith KA, Zalupski MM, Reese JB, Gearhart SL, Azad NS, Chan J, Olsen L, Efron JE, Lawrence TS, Ben-Josef E. The quality-of-life effects of neoadjuvant chemoradiation in locally advanced rectal cancer. Int J Radiat Oncol Biol Phys. 2013 Jan 1;85(1):e15-9. doi: 10.1016/j.ijrobp.2012.09.006. Epub 2012 Oct 9. PMID 23058059
- [Result] Pramateftakis MG, Kanellos D, Tekkis PP, Touroutoglou N, Kanellos I. Rectal cancer: multimodal treatment approach. Int J Surg Oncol. 2012;2012:279341. doi: 10.1155/2012/279341. Epub 2012 Sep 12. No abstract available. PMID 23008766
- [Result] Gillis C, Fenton TR, Sajobi TT, Minnella EM, Awasthi R, Loiselle SE, Liberman AS, Stein B, Charlebois P, Carli F. Trimodal prehabilitation for colorectal surgery attenuates post-surgical losses in lean body mass: A pooled analysis of randomized controlled trials. Clin Nutr. 2019 Jun;38(3):1053-1060. doi: 10.1016/j.clnu.2018.06.982. Epub 2018 Jul 9. PMID 30025745
- [Result] Wright S, Wiechula R, McLiesh P. The effectiveness of prehabilitation for adults having elective surgery: a systematic review protocol. JBI Database System Rev Implement Rep. 2016 Feb;14(2):78-92. doi: 10.11124/jbisrir-2016-2460. No abstract available. PMID 27536795
- [Result] Santa Mina D, van Rooijen SJ, Minnella EM, Alibhai SMH, Brahmbhatt P, Dalton SO, Gillis C, Grocott MPW, Howell D, Randall IM, Sabiston CM, Silver JK, Slooter G, West M, Jack S, Carli F. Multiphasic Prehabilitation Across the Cancer Continuum: A Narrative Review and Conceptual Framework. Front Oncol. 2021 Jan 11;10:598425. doi: 10.3389/fonc.2020.598425. eCollection 2020. PMID 33505914